CLINICAL TRIAL: NCT04512703
Title: Ambulatory Remote Patient Monitoring With the µCor Heart Failure and Arrhythmia Management System (PATCH) Feasibility Study
Brief Title: Feasibility Study of the µCor Heart Failure and Arrhythmia Management System (PATCH)
Acronym: PATCH
Status: Completed | Type: Observational
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 90D0167
Record Dates: First submitted 2020-07-31; First posted 2020-08-13 (Actual); Results first posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Heart Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (4):
- Healthy Group: Healthy male and female volunteers. Subjects older than 21 years of age. Subjects to wear the µCor device for up to 30 days.
  Interventions: Device: µCor
- Arrhythmia Monitoring Group: Patients with a clinical indication for outpatient cardiac monitoring. Subjects older than 21 years of age. Subjects to wear the µCor device for up to 90 days.
  Interventions: Device: µCor
- Front Position Devices: All devices placed in the front position
- Side Position Devices: All devices placed in the side position

INTERVENTIONS:
Device: µCor — Sensor Monitor for arrhythmia and other bio-metric markers
  Groups: Arrhythmia Monitoring Group; Healthy Group

SUMMARY:
Prospective, non-interventional, feasibility study. 8 months, from start of screening to finishing the study. Multi-center study, with a maximum of 8 centers in Europe. Health adult volunteers (21 years or older) and adult patients with a clinical indication for ambulatory outpatient cardiac monitoring.

To observe the feasibility of remotely monitoring patients with the novel µCor Heart Failure and Arrhythmia Management System (µCor system ) that non-invasively captures thoracic fluid content, electrocardiogram, heart rate, respiratory rate, activity, and body posture. tory outpatient cardiac monitoring.

DETAILED DESCRIPTION:
The study will consist of two phases. Phase I of the study will enroll 6 healthy volunteers, who have no indication for remote cardiac monitoring. Subjects are required to participate in the study for 30 days.

Phase II of the study will enroll up to 44 patients indicated for outpatient cardiac monitoring and will participate in the study for up to 90 days.

All subjects will wear the device in two locations, one along the left midaxillary line and the other along the left midclavicular line for the first seven days.

Thereafter, for the remainder of the study, half the enrolled subjects will only wear the device in the left midclavicular position and the other half will wear the device in the left midaxillary position. Subjects will use a diary to keep a daily log their activities of daily living (phase I) or a log of any symptoms related to heart rhythm abnormalities and heart failure (phase II).

Data will be acquired with the µCor system and wirelessly transmitted daily to a remote server for processing, generating thoracic fluid content, ECG, heart rate, respiration rate, activity, and posture measurements. Investigators will have access only to ECG data.

Study staff will make weekly phone calls to subjects and record any new clinically actionable events. Patients will have monthly office visits. At the end of 30 days (phase I) or 90 days (phase II), patients will end wear and will complete the study follow-up questionnaire.

The study will enroll a maximum of 50 subjects. Six healthy volunteers will be enrolled for phase I of the study. Remaining 44 subjects will be enrolled for phase II and will have an indication of outpatient cardiac monitoring.

ELIGIBILITY:
-Inclusion Criteria

The following criteria will be used to include subjects in phase I portion of the study:

* Healthy male and female volunteers.
* Subjects older than 21 years of age.
* Subjects willing to wear the µCor device for up to 30 days.
* Subjects willing to answer weekly phone calls from the study staff.

The following criteria will be used to include subjects in phase II portion of the study:

* Patients with a clinical indication for outpatient cardiac monitoring.
* Patients older than 21 years of age.
* Patients willing to wear the µCor device for up to 90 days.
* Patients willing to make monthly (30-, 60-, and 90-day) office visits during the study period.
* Patients willing to answer weekly phone calls regarding their health status.
* Exclusion Criteria:

The following criteria will be used to exclude subjects from phases I and II portions of the study:

* Subjects reporting or planning to be pregnant.
* Subjects with any cardiac implantable electronic devices, including loop recorders.
* Subjects with a wearable cardioverter defibrillator.
* Subjects with Holter monitors, wearable event recorders, and other mobile cardiac telemetry devices.
* Subjects with any skin condition that would prevent them from wearing the µCor system.
* Subjects who are non-ambulatory.
* Subjects without adequate cellular transmission access that would prevent data download from the µCor device.
* Subjects participating in another clinical study.
* Subjects unable to give informed consent.
* Employees of ZOLL or their family members.
* Subjects traveling during the study participation period that prevents planned office visits and weekly phone calls from the study coordinator.
* Subjects expected to undergo a planned MRI exam during the participation period.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers (21 years or older) and adult patients with a clinical indication for ambulatory outpatient cardiac monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2020-08-02 (Actual); Study Completion 2020-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mike Osz, Study Director — Zoll Medical Corporation
Locations (1):
- Medizinische Hochschule Hannover, Hanover, Germany

IPD SHARING:
Plan to Share IPD: Undecided
undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: An additional subject was enrolled beyond the protocol in the arrhythmia group.
Period: Within 7 Days From Start of Device Wear
Arm/Group | Healthy Group | Arrhythmia Monitoring Group
Started | 6 | 45
Wore Front Position | 6 | 45
Wore Side Position | 6 | 45
Completed | 6 | 45
Not Completed | 0 | 0
Period: Between 7th and 90th Day of Device Wear
Arm/Group | Healthy Group | Arrhythmia Monitoring Group
Started | 6 | 45
Wore Side Position Device | 3 | 23
Wore Front Position Device | 3 | 22
Completed | 6 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Group | Arrhythmia Monitoring Group | Total
Number analyzed (Participants) | 6 | 45 | 51
Age, Continuous [Mean (Full Range); unit: years] | 35 [25 to 56] | 61 [19 to 79] | 58 [19 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 23 | 26
  Male | 3 | 22 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 6 | 45 | 51

OUTCOME MEASURES:

1. Primary Outcome: Logistics of Study Device Setup and Monitoring
Description: Logistics will be assessed by the number of subjects successfully fitted with a device that was able to transmit data to the remote server. Device Setup
Time Frame: Period 1: Start of device wear at Day 0 to Day 7 and Period 2: Day 8 to 90
Population: All devices in both Healthy and Arrythmia Monitoring Group were assessed for setup at the beginning of Period 1. Monitoring assessment was assessed during both Period 1 and Period 2. There was a total of 51 side position devices and 51 front position devices.
Measure: Number; unit: count of participants
Groups:
- Front Position Devices: Devices placed in the front position
- Side Position Devices: Devices placed in the side position
Arm/Group | Front Position Devices | Side Position Devices
Number analyzed (Participants) | 51 | 51
count of participants
  Devices Assessed for Setup during Period 1 | 51 | 51
  Devices Assessed for Monitoring during Period 1 | 51 | 51
  Devices assessed for Monitoring during Period 2 | 22 | 23

2. Primary Outcome: Device Wear Time and Compliance
Description: Total number of days the device is worn at least once, in the devices indicated for long term wear in the heart arryhthmia group. These devices were worn during both Period 1 and Period 2, and the outcome measure was assessed irrespective of whether the device was being worn in Period 1 or Period 2.
Time Frame: Period 1: Start of device wear at Day 0 to Day 7 and Period 2: Day 8 to 90
Population: Devices on subjects in the arrythmia group that were allocated for 90 day wear were used in the assessment.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Front Position Devices | Side Position Devices
Number analyzed (Participants) | 22 | 23
Days | 68 (29) | 54 (36)

3. Primary Outcome: Subject's Ability to Accurately Place Device
Description: Subject Training will be assessed by measuring the incidence of correct device placement. Correct device placement was assessed irrespective of whether the device was being worn in Period 1 or Period 2.
Time Frame: Period 1: Start of device wear at Day 0 to Day 7 and Period 2: Day 8 to 90
Population: A position assessment and orientation placement was assessed for accuracy for all front and side devices.
Measure: Number; unit: percentage of correct placements
Arm/Group | Front Position Devices | Side Position Devices
Number analyzed (Participants) | 51 | 51
percentage of correct placements | 96 | 96

4. Primary Outcome: Device Data Transmission and Device Connectivity
Description: Count of subjects that had daily data transmission.
Time Frame: Period 1 and Period 2
Measure: Number; unit: count of participants
Arm/Group | Front Position Devices | Side Position Devices
Number analyzed (Participants) | 51 | 51
count of participants
  Devices Worn during Phase 1 | 51 | 51
  Devices Worn during Phase 2 | 22 | 23

5. Primary Outcome: Ability to Provide Timely Arrythmia Monitoring
Description: Timely arrythmia monitoring will be assessed by the mean time from arrythmia event trigger to publication of arrythmia report to investigator. Timing or arrhythmia monitoring reporting was assessed irrespective of whether the device was being worn in Period 1 or Period 2.
Time Frame: Period 1: Start of device wear at Day 0 to Day 7 and Period 2: Day 8 to 90
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Front Position Devices: Devices placed in the front position indicated for 90 day monitoring
- Side Position Devices: Devices placed in the side position indicated for long term monitoring
Arm/Group | Front Position Devices | Side Position Devices
Number analyzed (Participants) | 22 | 23
hours | 9.9 (42.8) | 10.5 (55.0)

6. Primary Outcome: Documentation of Clinically Actionable Events.
Description: Assessed by the total number of clinical events documented including arrythmia symptoms, physician office visits, ER visits, hospitalizations, and mortality in both the healthy group and arrhythmia monitoring group. The number or clinical events documented was assessed irrespective of whether the device was being worn in Period 1 or Period 2.
Time Frame: Period 1: Start of device wear at Day 0 to Day 7 and Period 2: Day 8 to 90
Measure: Number; unit: documented clinical events
Arm/Group | Front Position Devices | Side Position Devices
Number analyzed (Participants) | 51 | 51
documented clinical events | 29 | 42

7. Secondary Outcome: Thoracic Fluid Content (TFC) Front and Side Device Measurement Equivalency
Description: The TFC measurement was compared between front and side placed devices. TFC is a unitless measurement that encompasses the degree of reflected radar waves in the lung taken by the study device. Higher TFC is indicative of increased fluid, whereas lower TFC is indicative of decreased fluid.
Time Frame: Period 1: Start of device wear at Day 0 to Day 7
Population: Includes both healthy and arrhythmia monitoring groups
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Front Position Devices | Side Position Devices
Number analyzed (Participants) | 51 | 51
units | 23.4 (7.3) | 24.0 (9.5)

8. Secondary Outcome: Association of Device Recordings to Clinical Events
Description: Device recordings were assessed and compared to clinical events in both the healthy group and arrhythmia monitoring group. Device recording associations were assessed irrespective of whether the device was being worn in Period 1 or Period 2.
Time Frame: Period 1: Start of device wear at Day 0 to Day 7 and Period 2: Day 8 to 90
Population: Devices in all subjects were assessed for arrythmia/symptom associations. The healthy and arrhthmia monitoring groups were combined for this outcome measure as the study investigated whether documented symptoms were associated with ECG arrhythmia regardless of group allocation.
Measure: Number; unit: Arrhythmias associated with symptoms
Groups:
- All Subjects: ECG arrythmia recordings were assessed for associations with documented symptoms in cases of arrhythmia reported symptoms
Arm/Group | All Subjects
Number analyzed (Participants) | 51
Arrhythmias associated with symptoms | 5

9. Secondary Outcome: Device Recording Stability
Description: Device recording stability was assessed through the heart rate coefficient of variation in both front and side placed devices. Stability was assessed irrespective of whether the device was being worn in Period 1 or Period 2.
Time Frame: Period 1: Start of device wear at Day 0 to Day 7 and Period 2: Day 8 to 90
Population: Includes both healthy and arrhythmia monitoring groups
Measure: Mean (Standard Deviation); unit: Percent Coefficient of Variation
Arm/Group | Front Position Devices | Side Position Devices
Number analyzed (Participants) | 51 | 51
Percent Coefficient of Variation | 0.48 (.47) | 0.41 (.20)

10. Secondary Outcome: Respiration Rate Front and Side Device Measurement Equivalency
Description: Respiration rates were compared between front and side placed devices. The outcome was measured only during Period 1 when both front and side devices were worn simultaneously.
Time Frame: Period 1: Start of device wear at Day 0 to Day 7
Population: Includes both healthy and arrhythmia monitoring groups
Measure: Mean (Standard Deviation); unit: respirations per minute
Arm/Group | Front Position Devices | Side Position Devices
Number analyzed (Participants) | 51 | 51
respirations per minute | 16.9 (4.4) | 16.9 (4.4)

11. Secondary Outcome: Activity Front and Side Device Measurement Equivalency
Description: Activity counts were compared between front and side devices.
Time Frame: Period 1: Start of device wear at Day 0 to Day 7
Population: Includes both healthy and arrhythmia monitoring groups
Measure: Mean (Standard Deviation); unit: activity counts
Arm/Group | Front Position Devices | Side Position Devices
Number analyzed (Participants) | 51 | 51
activity counts | 981 (934) | 1007 (989)

12. Secondary Outcome: Sleep Angle Front and Side Device Measurement Equivalency
Description: Sleep angle was compared between front and side devices.
Time Frame: Period 1: Start of device wear at Day 0 to Day 7
Population: Includes both healthy and arrhythmia monitoring groups
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Front Position Devices | Side Position Devices
Number analyzed (Participants) | 51 | 51
degrees | 2.5 (12.8) | 2.3 (12.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment of the subject in the study to the date the subject completed the study, up to 90 days.
Description: Adverse evenst were defined in the study as any untoward medical occurrence, unintended disease or injury or any untoward clinical signs in subjects, users, or other persons whether or not related to the study device.
  Serious adverse events were defined per study protocol.
Arm/Group | Healthy Group | Arrhythmia Monitoring Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/45
Other Adverse Events (participants affected / at risk) | 6/6 | 42/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Group (N=6) | Arrhythmia Monitoring Group (N=45)
Skin Irritation (Skin and subcutaneous tissue disorders) | 6 | 42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any proposed publication relating to the research conducted under this protocol will be submitted to the sponsor for review at least 45 days prior to submission for publication. The publication may be delayed for an additional period of up to 90 days for intellectual property considerations or until all confidential information has been eliminated from the publication(s) and sponsor has approved the publication. It may be determined by the sponsor that no data from this study will be published.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/03/NCT04512703/Prot_SAP_000.pdf